CLINICAL TRIAL: NCT04843943
Title: An Exploratory Study of Sintilimab in Combination With Bevacizumab Biosimilar in Patients With Potentially Resectable Intermediate HCC
Brief Title: Sintilimab Combined With Bevacizumab Biosimilar for Potentially Resectable Intermediate HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jia Fan, Director of hospital, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-156(2)R
Record Dates: First submitted 2021-04-08; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Bevacizumab (Experimental)
  Interventions: Drug: Sintilimab; Drug: Bevacizumab Biosimilar

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: 200mg IV Q3W D1
Drug: Bevacizumab Biosimilar — Bevacizumab biosimilar: 15mg/kg, IV, Q3W, D1

SUMMARY:
This is a Phase Ib study to evaluate the safety and efficacy of sintilimab combined with bevacizumab biosimilar in patients with potentially resectable intermediate hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent and willing to sign an approved consent form
2. Age 18-75, male and female
3. Potentially resectable Intermediate (CNLC-IIa and IIb) HCC with diagnosis confirmed by histology/cytology or clinically
4. No prior therapy for HCC
5. Child-Pugh: A
6. ECOG PS: 0-1
7. Expected survival ≥6 months
8. Measurable disease per RECIST1.1
9. Major organ functions meet the following requirements:

   no blood transfusion, no use of hematopoietic stimulators (including g-csf, gm-csf, EPO and TPO) and infusion of human albumin preparations within 14 days prior to screening: neutrophil absolute count ≥1.0×10^9/L;Platelet count ≥ 75×10^9/L;Hemoglobin ≥ 9 g/dL;Serum albumin ≥ 2.8 g/dL;Total serum bilirubin ≤2.0× upper limit of normal range (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN;Serum creatinine (Cr) ≤1.5×ULN or Cr clearance ≥30 mL/min (calculated by Cockcroft-Gault formula);International standardized ratio (INR) ≤1.5×ULN;
10. Women of childbearing age must undergo a blood pregnancy test within the first 3 days of randomization with negative results and agree to use a reliable and effective method of contraception during the trial and within 120 days of the last trial drug administration. Male patients whose partners are women of childbearing age must agree to use a reliable and effective method of contraception during the trial and within 120 days of the last trial drug administration.

Exclusion Criteria:

1. known as cholangiocarcinoma (ICC) or mixed hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and hepatic fibrolamellar carcinoma.
2. History of organ transplantation or hepatic encephalopathy
3. Tumor accumulation range exceeds 70% of liver volume
4. Pleural fluid, ascites, and pericardial effusion with clinical symptoms requiring drainage
5. Any history of kidney disease or nephrotic syndrome
6. History of gastrointestinal (GI) perforation and/or fistula in the past 6 months;Severe (G3) varicose veins are known to be present on endoscopy within 3 months before the first dose ; history of thrombosis, bleeding diathesis, coagulopathy or significant vascular disease
7. Prior life-threatening blood loss or grade 3/4 gastrointestinal bleeding requiring blood infusion, endoscopic or surgical intervention within 3 months
8. Arterial and venous thromboembolic events in the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other serious thromboembolism history.
9. Severe bleeding tendency or coagulopathy, or are receiving thrombolytic therapy
10. Long-term use of vitamin K antagonists (such as warfarin) or low-dose low-molecular-weight heparin (such as enoxaparin 40 mg/day) or heparin
11. Uncontrollable hypertension, systolic blood pressure> 140 mmHg or diastolic blood pressure> 90 mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy
12. Symptomatic congestive heart failure (New York Heart Association Grade II-IV), symptomatic or poorly controlled arrhythmia, history of congenital long QT syndrome or QTc> 500ms corrected during screening
13. History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months of initiation of study treatment
14. Had major surgical procedure within 4 weeks of initiation of study treatment
15. Past and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severely impaired lung function and other lung diseases
16. Had acute or chronic active hepatitis B or C infection. Hepatitis C virus (HCV) RNA>103 copies/ml; hepatitis B surface antigen (HbsAg) and anti-HCV antibody are positive at the same time; hepatitis B virus (HBV) DNA positive but has received antiviral treatment is allowed.
17. Had active tuberculosis (TB)
18. Had human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive), known syphilis infection
19. Had severe infections that are active or poorly clinically controlled.
20. Had active autoimmune disease
21. Have used immunosuppressive drugs within 4 weeks before the first dose
22. Received live attenuated vaccines within 4 weeks before the first dose or plan to receive live attenuated vaccines during the study period
23. Received Chinese medicine with anti-tumor indications, or received drugs with immunomodulatory effect within 2 weeks before the first administration
24. Received any anti-PD-1 antibody, anti-PD-L1/L2 antibody, anti-CTLA4 antibody, or other immunotherapy
25. Allergic to Sintilizumab, Bevacizumab preparations and excipients, or had severe allergic reactions to other monoclonal antibodies in the past
26. Received treatment from other clinical trials within 4 weeks before the first dose
27. Female patients who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 2 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0; Surgical safety including Intraoperative blood loss，PHLF assessed by ISGLS（2012），Postoperative complications evaluated by modified Clavien-Dindo system
Events Free Survival (EFS) Assessed by RECIST1.1 | Up to 2 years
  Defined as the time from enrollment to disease progression, recurrence or death (whichever occurs first)

SECONDARY OUTCOMES:
resection rate (R0 resection rate) | Up to 2 years
  Defined as the proportion of patients undergoing radical resection to the total subjects (R0 resection rate)
Pathological response rate | Up to 2 years
  Defined as the proportion of patients who had pathological response.
Objective response rate (ORR) assessed by RECIST1.1 | Up to 2 years
  Defined as the proportion of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR).
Recurrence-free survival (RFS) of patients who accepted surgery | Up to 2 years
  Defined as the time from the date of surgery to the date of disease recurrence or death whichever occur first, assessed up to 2 years post-treatment
Progression free survival (PFS) assessed by RECIST1.1 of patients who didn't accept surgery | Up to 2 years
  Defined as the time from initiation of treatment until the first occurrence of disease progression or death from any cause, whichever occurs first.
Overall survival (OS) of the patients who accepted surgery | Up to 2 years
  Defined as the time from the date of treatment start to the date of death or to the date of last follow-up for patients alive.
Overall survival (OS) of the patients who didn't accepted surgery | Up to 2 years
  Defined as the time from the date of treatment start to the date of death or to the date of last follow-up for patients alive.
Overall survival (OS) | Up to 2 years
  Defined as the time from the date of treatment start to the date of death or to the date of last follow-up for patients alive

REFERENCES:
- [Derived] Sun HC, Zhu XD, Wang ZY, Gao Q, Ji Y, Shi YH, Wang XY, Qiu SJ, Huang C, Shen YH, Zhou J, Fan J. Sintilimab plus bevacizumab followed by resection in intermediate-stage hepatocellular carcinoma: a phase Ib clinical trial with biomarker analysis. BMJ Oncol. 2024 Dec 16;3(1):e000578. doi: 10.1136/bmjonc-2024-000578. eCollection 2024. PMID 40046248